CLINICAL TRIAL: NCT06411574
Title: Comparing the Impact of Body Surface Gastric Mapping and Gastric Emptying Scintigraphy on Clinical Management in Suspected Gastroparesis
Brief Title: Body Surface Gastric Mapping Vs Gastric Emptying Scintigraphy on Clinical Management in Gastroparesis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Western Sydney (Other)
Collaborators: University of Auckland, New Zealand (Other)
Responsible Party: Principal Investigator, Vincent Ho, Associate Professor, University of Western Sydney
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: WS-GMSC-001
Record Dates: First submitted 2024-04-28; First posted 2024-05-13 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2024-12

CONDITIONS: Gastroparesis
Keywords: Gastroparesis; Motility Disorders; Gastric Emptying Scintigraphy; Body Surface Gastric Mapping
MeSH Terms: conditions — Gastroparesis

STUDY DESIGN:
Intervention Model Description: Participants will be recruited into one of two groups: standard of care (GES only) or BSGM-guided care (GES + BSGM). Each group will undergo treatment based on their respective management plan.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of care (No Intervention): Only the GES test result will be used to guide treatment as part of standard of care.
- BSGM-guided care (Experimental): Both the GES and BSGM test results will be used to guide treatment.
  Interventions: Device: Gastric Alimetry

INTERVENTIONS:
Device: Gastric Alimetry — The Gastric Alimetry™ System is intended to record, store, view and process gastric myoelectrical activity as an aid in the diagnosis of various gastric disorders.
  Arms: BSGM-guided care

SUMMARY:
Gastroparesis is a chronic and debilitating gastric disease associated with poor quality of life, psychological distress, frequent hospitalisations, and high healthcare utilization and associated costs. It is defined by persistent upper gastrointestinal symptoms and delayed gastric emptying with no mechanical gastric outlet obstruction. Gastric emptying scintigraphy (GES) is the current gold standard for diagnosing gastroparesis but its clinical utility is currently being questioned. Current management strategies have often been found to be ineffective, largely due to an incomplete understanding of the disease's pathophysiology. There is a critical need for more advanced diagnostic testing that can better diagnose patients and guide personalized targeted therapy.

Body surface gastric mapping (BSGM) using Gastric Alimetry (Alimetry Ltd., New Zealand) is a new FDA-cleared medical device to assess gastric function by non-invasively assessing gastric motility using simultaneous high-resolution electrogastrography and symptom profiling. BSGM has demonstrated clinical utility in the assessment of gastric function through patient phenotyping in a variety of cohorts, including patients with nausea and vomiting disorders, diabetes, delayed gastric emptying, and post-gastric surgery. Previous research revealed that the detection of gastric motility abnormality rates through patient phenotyping were higher using Gastric Alimetry compared to GES (43% vs 23%). Clinical application of these phenotypes has also aided in changing management decisions, which reduced healthcare utilization and associated costs. However, how GES and BSGM test results differentially influence clinical management in patients is uncertain.

This exploratory pilot study proposes a two-arm, prospective trial to assess whether BSGM-guided care could change clinical outcomes compared to the standard of care (GES) in patients with suspected gastroparesis. The trial consists of two phases. Phase 1 involves participants separately undertaking a GES and BSGM test. Based on these results, the referring clinician will devise management plans for treatment using a standardized form: 1) unblinded to one test (GES or BSGM) but blinded to the other test; and 2) unblinded to both tests (GES + BSGM). They will be asked to recommend any changes to interventions (medications, diet, endoscopic/surgical referral or other) and additional testing. In phase 2, those in Phase 1 will undergo BSGM-guided care based on their combined management plan (GES + BSGM) and followed up over a 12 month period. A separate set of participants will be recruited to undergo standard of care (GES only) in parallel with Phase 1 participants. After 12 months, those on the standard of care arm will be crossed over to BSGM-guided care, undergo a BSGM test, treated according to the new management plan, and followed up over 6 months. Questionnaires will assess symptoms, quality of life, health psychology, sleep, and work impact.

If validated, this may change clinical practice by reducing the need for invasive or radioactive-based procedures to diagnose these patients and facilitating a more targeted treatment approach.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 18 years old
* Meeting Rome IV Criteria for Functional Dyspepsia and/or Chronic Nausea and Vomiting Syndrome
* Referred for gastric emptying scintigraphy
* Normal gastroscopy
* Negative or treated H. Pylori status

Exclusion Criteria:

* Pregnant or breast-feeding
* Inability to perform a BSGM test according to Indications for Use: history of severe skin allergies or sensitivity to cosmetics or lotions; chronically damaged or vulnerable epigastric skin (fragile skin, wounds, inflammation); unable to remain in a relaxed reclined position for the test duration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-05-03 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-12-03 (Estimated)

PRIMARY OUTCOMES:
Change in clinical management decisions based on the combined test results. | Baseline
  A change constitutes any change within a category (e.g. from a prokinetic to neuromodulator, from one prokinetic to another), addition of category or removal of category. If the plan remains the same, this is considered no change.
Healthcare utilization (expressed as work impairment percentages; higher scores meaning worse outcome) between standard of care and BSGM-guided care. | 12 months.
  Work impairment scale is Work Productivity and Activity Impairment Questionnaire: General Health V2.0 (minimum: 0; maximum: 100).
Healthcare utilization-associated costs (expressed as the total amount in AUD) between standard of care and BSGM-guided care. | 12 months.
  Costs associated with healthcare events (emergency department visits, hospital admissions, gastroenterology clinic visits and investigations) before and after testing.

SECONDARY OUTCOMES:
Change in clinical management decisions based on order of unblinding motility test results (GES then BSGM vs BSGM then GES). | Baseline
  A change constitutes any change within a category (e.g. from a prokinetic to neuromodulator, from one prokinetic to another), addition of category or removal of category. If the plan remains the same, this is considered no change. The change will then be compared between unblinding GES then BSGM vs BSGM then GES.
Change in Gastroparesis Cardinal Symptom Index (minimum: 0; maximum: 5) scores between standard of care and BSGM-guided care (with a higher score meaning worse outcome). | 12 months.
Change in Patient Assessment of Upper Gastrointestinal Symptom Severity Index (minimum: 0; maximum: 5) scores between standard of care and BSGM-guided care (with a higher score meaning worse outcome). | 12 months.
Change in Patient Assessment of Upper GastroIntestinal Disorders-Quality of Life (minimum: 0; maximum: 5) scores between standard of care and BSGM-guided care (with a lower score meaning worse outcome). | 12 months.
Change in 5-level EQ-5D (minimum: 0; maximum: 1) scores between standard of care and BSGM-guided care (with a lower score meaning worse outcome). | 12 months.
Change in Patient Health Questionnaire-8 (minimum: 0; maximum: 24) scores between standard of care and BSGM-guided care (with a higher score meaning worse outcome). | 12 months.
Change in General Anxiety Disorder-7 (minimum: 0; maximum: 21) scores between standard of care and BSGM-guided care (with a higher score meaning worse outcome). | 12 months.
Change in Perceived Stress Scale-4 (minimum: 0; maximum: 4) scores between standard of care and BSGM-guided care (with a higher score meaning worse outcome). | 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Ho, MBBS, FRACP, FACP, PhD, Principal Investigator — Western Sydney University
Locations (1):
- Western Sydney University, Campbelltown, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gharibans AA, Calder S, Varghese C, Waite S, Schamberg G, Daker C, Du P, Alighaleh S, Carson D, Woodhead J, Farrugia G, Windsor JA, Andrews CN, O'Grady G. Gastric dysfunction in patients with chronic nausea and vomiting syndromes defined by a noninvasive gastric mapping device. Sci Transl Med. 2022 Sep 21;14(663):eabq3544. doi: 10.1126/scitranslmed.abq3544. Epub 2022 Sep 21. PMID 36130019
- [Background] Varghese C, Schamberg G, Calder S, Waite S, Carson D, Foong D, Wang WJ, Ho V, Woodhead J, Daker C, Xu W, Du P, Abell TL, Parkman HP, Tack J, Andrews CN, O'Grady G, Gharibans AA. Normative Values for Body Surface Gastric Mapping Evaluations of Gastric Motility Using Gastric Alimetry: Spectral Analysis. Am J Gastroenterol. 2023 Jun 1;118(6):1047-1057. doi: 10.14309/ajg.0000000000002077. Epub 2022 Dec 20. PMID 36534985
- [Background] Wang WJ, Foong D, Calder S, Schamberg G, Varghese C, Tack J, Xu W, Daker C, Carson D, Waite S, Hayes T, Du P, Abell TL, Parkman HP, Huang IH, Fernandes V, Andrews CN, Gharibans AA, Ho V, O'Grady G. Gastric Alimetry Expands Patient Phenotyping in Gastroduodenal Disorders Compared with Gastric Emptying Scintigraphy. Am J Gastroenterol. 2024 Feb 1;119(2):331-341. doi: 10.14309/ajg.0000000000002528. Epub 2023 Oct 30. PMID 37782524
- [Background] Varghese C, Daker C, Lim A, Sebaratnam G, Xu W, Kean B, Cederwall C. Gastric Alimetry in the Management of Chronic Gastroduodenal Disorders: Impact to Diagnosis and Health Care Utilization. Clin Transl Gastroenterol. 2023 Nov 1;14(11):e00626. doi: 10.14309/ctg.0000000000000626. PMID 37589479
- [Background] Varghese C, Xu W, Daker C, Bissett IP, Cederwall C. Clinical utility of Gastric Alimetry® in the management of intestinal failure patients with possible underlying gut motility disorders. Clinical Nutrition Open Science [Internet]. 2023 Oct 1;51:15-25. Available from: https://www.sciencedirect.com/science/article/pii/S2667268523000359.
- [Background] Xu W, Gharibans AA, Calder S, Schamberg G, Walters A, Jang J, Varghese C, Carson D, Daker C, Waite S, Andrews CN, Cundy T, O'Grady G. Defining and Phenotyping Gastric Abnormalities in Long-Term Type 1 Diabetes Using a Novel Body Surface Gastric Mapping Device. Gastro Hep Adv. 2023 Aug 18;2(8):1120-1132. doi: 10.1016/j.gastha.2023.08.005. eCollection 2023. PMID 39131562
- [Background] Xu W, Wang T, Foong D, Schamberg G, Evennett N, Beban G, Gharibans A, Calder S, Daker C, Ho V, O'Grady G. Characterization of gastric dysfunction after fundoplication using body surface gastric mapping. J Gastrointest Surg. 2024 Mar;28(3):236-245. doi: 10.1016/j.gassur.2023.12.023. Epub 2024 Jan 23. PMID 38445915